CLINICAL TRIAL: NCT06874192
Title: Safety and Efficacy of LOw DOse COlchicine in Patients With STatin INTolerance: the LODOCO STINT Pilot Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20030934
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Statin Adverse Reaction
Keywords: statin intolerance

STUDY DESIGN:
Intervention Model Description: Single-center, double-blind, placebo-controlled, randomized cross-over pilot study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomized in a 1:1 ratio to receive either low-dose colchicine (0.5 mg once daily) or matching placebo for 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose colchicine and then matching placebo (Experimental): Participants in this arm will be randomized to receive low-dose colchicine (0.5 mg once daily) and then placebo for 4 weeks
  Interventions: Drug: Low-dose colchicine at 0.5mg daily; Other: Placebo
- Matching placebo and then low dose colchicine (Experimental): Participants in this arm will be randomized to receive placebo for 4 weeks and then low-dose colchicine (0.5 mg once daily)
  Interventions: Drug: Low-dose colchicine at 0.5mg daily; Other: Placebo

INTERVENTIONS:
Drug: Low-dose colchicine at 0.5mg daily — LODOCO is low-dose colchicine at 0.5mg daily, ii is an FDA approved anti-inflammatory drug, to prevent cardiovascular events in patients with coronary artery disease. LODOCO works by inhibiting microtubule formation and reducing the activity of neutrophils, which play a key role in inflammation.
Other: Placebo — Matching placebo

SUMMARY:
Statins are a class of cholesterol lowering medications that contribute to reducing a person's risk of experiencing a cardiovascular event like heart attack. Along with the ability to lower cholesterol, statins also possess anti-inflammatory properties which contribute to their cardioprotective effects. Some people experience side effects while taking statins and are unable to continue treatment with them,which can then increase a person's risk of having cardiovascular issues due to untreated high cholesterol levels. Prior studies have shown that inflammation in the body may lead to an increased risk of a future cardiovascular events. Low dose colchicine (LODOCO), an anti-inflammatory agent, has been shown to reduce cardiovascular events by inhibiting inflammation, a major cause of cardiovascular disease. The United States Food and Drug Administration (FDA) has approved LODOCO to reduce the risk of a future cardiac events for those who have existing heart disease or possess multiple risk factors for heart disease.

DETAILED DESCRIPTION:
This study will test the effects of LODOCO in those who have previously been identified as statin intolerant, meaning they are unable to continue taking statins because of side effects. The primary objective of this study is to evaluate the safety and efficacy of low-dose colchicine (LODOCO) in subjects with statin intolerance. Safety will be assessed by monitoring the incidence of adverse events from baseline to four weeks. Efficacy will be determined by measuring the change in high-sensitivity C-reactive protein (hs-CRP) levels from baseline to four weeks..

ELIGIBILITY:
Inclusion Criteria:

* History of statin intolerance (As defined by the NLA 2023 guidelines) Patients who have experienced one or more adverse effects associated with statin therapy, which resolves or improves with dose continuation or reduction
* Stable dose of lipid-lowering regimen (statin or non-statin) for at least one month
* Patients able to provide informed consent.
* Aged 18 to 80 will be enrolled in the study.

Exclusion Criteria:

* Known hypersensitivity to colchicine, current use of colchicine or other anti-inflammatory medications.
* Renal impairment (eGFR <45 mL/min/1.73 m2)
* Transaminitis (ALT or AST >3 times upper limit of normal)
* Cirrhosis
* Severe Heart Failure
* Active cancer or currently on chemotherapy
* Irritable Bowel Syndrome, Inflammatory Bowel Disease (Crohn's or Ulcerative Colitis) or other diarrheal related GI pathologies
* Active infection
* Autoimmune or inflammatory condition
* Pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety will be assessed by monitoring the incidence of adverse events | Baseline to four weeks.
  Safety will be assessed by monitoring the incidence of adverse events from baseline to four weeks. Adverse events and tolerability will be evaluated using investigator-administered questionnaires at scheduled study visits. Participants will be asked to self-report any symptoms between visits, and all adverse events will be documented.
Efficacy will be determined by measuring the change in high-sensitivity C-reactive protein | Baseline to four weeks
  Efficacy will be determined by measuring the change in high-sensitivity C-reactive protein (hs-CRP) levels from baseline to four weeks. The measurement of hs-CRP pre and post treatment will assess the change in hs-CRP with colchicine. This will test the hypothesis that LODOCO through the inhibition of the inflammatory pathways will lead to a decrease in hs-CRP levels.

SECONDARY OUTCOMES:
To investigate the changes in interleukin-6 (IL-6) levels with low-dose colchicine therapy in patients with statin intolerance. | baseline to four weeks
  To assess the impact of low dose colchicine on IL-6, we will measure serum IL-6 levels in patients with statin intolerance at baseline and after 30 days of low-dose colchicine therapy. We hypothesize that there will be a significant reduction in IL-6 levels, reflecting a decrease in systemic inflammation.
To assess changes in lipid profile from baseline to 30 days | baseline to four weeks.
  To evaluate lipid profile changes in statin-intolerant patients receiving low-dose colchicine by measuring total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), triglycerides, low-density lipoprotein cholesterol (LDL-C), and lipoprotein(a) [Lp(a)] at baseline and after 30 days of therapy. A 30-day time frame allows for observation of early changes in lipid parameters, which may help guide longer-term studies and inform clinical decision-making.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Mehta, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No